CLINICAL TRIAL: NCT01144351
Title: A Phase 1b, Dose-Escalating, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety and Efficacy of Subcutaneous ELND002 in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: A Safety and Efficacy Study of ELND002 in Patients With Relapsing Forms of Multiple Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELND002-MS103
Record Dates: First submitted 2010-06-09; First posted 2010-06-15 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
Keywords: MS; SPMS; RRMS; Relapsing Forms of Secondary Progressive Multiple Sclerosis (SPMS); or Relapsing-Remitting Multiple Sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ELND002 (Experimental): ELND002 sc injection
  Interventions: Drug: ELND002
- Placebo (Placebo Comparator): placebo injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ELND002
  Arms: ELND002
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of ELND002 in patients with relapsing forms of secondary progressive multiple sclerosis (SPMS) or relapsing-remitting multiple sclerosis (RRMS).

ELIGIBILITY:
Inclusion Criteria:

* Has either clinically definite or laboratory-supported definite relapsing forms of MS for at least 2 years
* Patients with SPMS or RRMS have documented medical history of relapse in the past year or MRI-documented evidence of MS activity in the past year
* Has had an inadequate response or intolerability to interferon and/or glatiramer acetate
* Is able and willing to undergo Gd administration and repeat MRI testing

Exclusion Criteria:

* Has primary progressive MS (PPMS)
* Any history of treatment with recombinant humanized monoclonal antibodies
* Has received treatment with immunosuppressant medications or experimental agents within 3 months prior to the Baseline
* A history of opportunistic infection or the presence of any active infection within 3 months prior to Baseline
* Any history of congestive heart failure or currently has a pacemaker
* Has a known or suspected hypersensitivity to sulfonamides or any of the components of the investigational drug
* Has any medical history or psychiatric condition that would impact outcome or study participation
* Has other clinically significant abnormality on physical, neurological, laboratory, or ECG examination as listed in the protocol during the Screening Phase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of ELND002 including the identification of dose-limiting toxicity(ies) (DLT) and determination of the maximum tolerated dose (MTD) in patients with multiple sclerosis (MS). | 12 weeks

SECONDARY OUTCOMES:
Assessment of PK and PD measures of ELND002 (including but not limited to Cmax, Tmax, T1/2, AUC) | 12 weeks
  Measurement of drug concentration, alpha 4 receptor saturation, soluble VCAM and MADCAM.
Assessment of the cumulative number and volume of Gd-enhancing T1-weighed MRI brain lesions | 12 weeks
Reduction in rate of clinical relapses. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- United States (17):
  - Research Site, Berkeley, California
  - Research Site, Fresno, California
  - Research Site, Newport Beach, California
  - Research Site, Aurora, Colorado
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Northbrook, Illinois
  - Research Site, Farmington Hills, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Albuquerque, New Mexico
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Uniontown, Ohio
  - Research Site, Cordova, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec